CLINICAL TRIAL: NCT05265468
Title: Noninvasive Treatment of Upper Trapezius Active Trigger Points in College Students With Neck Pain. A Randomized Clinical Trial
Brief Title: Noninvasive Treatment of Upper Trapezius Active Trigger Points in College Students With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Juan Martínez Fuentes, Study Director, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE112103
Record Dates: First submitted 2022-01-20; First posted 2022-03-03 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Neck Pain; Trigger Point Pain, Myofascial
Keywords: Physiotherapy; Rehabilitation; Treatment; Active Trigger Point
MeSH Terms: conditions — Neck Pain; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Jones Group (Strain Counterstrain) (Experimental): Jones Group consist in 90 seconds in a ralease positioning of no pain in muscle acortation
  Interventions: Other: Jones Group (Strain Counterstrain)
- Lewit Group (Active Comparator): Lewit Group consist in a maximum of four minutes of muscular contraction acompaind by stretching techniques
  Interventions: Other: Lewit Group
- Chaitow Group (Active Comparator): Chaitow Group consist in a maximum of four minutes of muscular contraction acompaind by stretching techniques and deep diaphragmatic respiration
  Interventions: Other: Chaitow Group
- Placebo Group (Placebo Comparator): Placebo Group only have to mantain no pain positioning for 3 minutes
  Interventions: Other: Placebo Group

INTERVENTIONS:
Other: Jones Group (Strain Counterstrain) — No pain positioning technique with diaphragmatic breathing
  Arms: Jones Group (Strain Counterstrain)
Other: Lewit Group — Isometric muscular exercise acompained with stretching technique
  Arms: Lewit Group
Other: Chaitow Group — Isometric muscular exercise acompained with stretching technique and diaphragmatic breathing
  Arms: Chaitow Group
Other: Placebo Group — No pain positioning of participants
  Arms: Placebo Group

SUMMARY:
Hyperexcitable myofascial trigger points located within a taut band of skeletal muscle or fascia cause referred pain, local tenderness, and autonomic changes. The scientific data refer to an immediate improvement in the symptoms of these active points treated with manual therapy. Based on these factors, the objective of the study is to determine the effect of the combined therapy of the Jones, Chaitow, Lewit technique and pain-free positioning in participants with the presence of an active upper trapezius trigger point.

DETAILED DESCRIPTION:
The treatment will last a total of 15 minutes accompanied by a baseline assessment and after 10 minutes of the intervention in 3 experimental groups and a placebo group, of no-pain positioning. In addition to basic indices and scales of cervical pain and functionality, it is intended to measure flexibility, range of motion, proprioception and cognition through software with sensors of the latest technology when it comes to representing reliable results in differences between techniques.

ELIGIBILITY:
Inclusion Criteria:

* persistent neck pain or headache for more than 3 days
* presence of active trigger point in upper trapezius

Exclusion Criteria:

* Participants who present dizziness, vertigo and/or symptoms aggravated by the movement and/or positioning of the neck;
* who present infection or febrile state at the time of performing the test;
* with anxiety and/or extreme emotional tension;
* who are undergoing pharmacological treatment (analgesics, muscle relaxants, anxiolytics, antidepressants)

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 10 minutes
  Self-completed neck questionnaire wich consists in 10 sections. Each one of them (cervical pain intensity, personal care, lifting weights, reading, headache, ability to concentrate, ability to work, driving, sleep and leisure activities) offers 6 possible answers that represent 6 progressive levels of functional capacity, and is scored from 0 to 5. The total score is expressed in percentage terms with respect to the maximum possible
Pain intensity | 10 minutes
  Measured with Numeric Rating Scale wich consist in measure pain intensity with a score of 0-10
Pression algometer | 10 minutes
  Measures pressure pain thresholds

SECONDARY OUTCOMES:
Cervical Test | 10 minutes
  Measured with Baiobit Software. The range of movement will be measured in grades as per: flexion/extension; right/left rotation; and right/left inclination
Proprioceptive Test | 10 minutes
  Measured with Baiobit Software o'clock test in a high/medium/low levels wich consist in a velocity and accuracy evaluation of combined cervical movements in the o'clock game test.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Murcia, Murcia, Spain